CLINICAL TRIAL: NCT00791713
Title: A Randomized, Open-label, Single-center, Crossover Study of the Potential Effects of Paroxetine on the Pharmacokinetics of a Single Dose of Paliperidone Extended-release in Healthy Men
Brief Title: A Study of the Effects of Paroxetine on the Pharmacokinetics of Paliperidone ER
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR007561
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2009-01

CONDITIONS: Schizophrenia
Keywords: Paliperidone ER; Antipsychotic drugs; Selective serotonin reuptake inhibitors; Mood disorders; Schizophrenia
MeSH Terms: conditions — Schizophrenia; Mood Disorders | interventions — Paliperidone Palmitate

INTERVENTIONS:
Drug: Paliperidone ER

SUMMARY:
The purpose of this study is to evaluate the effects of a CYP2D6 inhibitor, paroxetine, on the pharmacokinetics of a single dose of orally administered paliperidone ER and to evaluate the safety and tolerability of both treatments in healthy men

DETAILED DESCRIPTION:
This is a randomized, open-label, single-center, single-dose, 2 treatment, 2 way crossover study. It consists of 3 phases: a screening phase beginning within 21 days before the first study drug administration; an open label treatment phase consisting of 2 treatment periods (Period 1 and Period 2), during which patients will receive 2 single doses of 3 mg paliperidone ER; and end of study evaluations upon completion of all the study procedures in Period 2 or at early withdrawal. All volunteers will receive each of the following 2 treatments in random order: Treatment A: 1 tablet of 3 mg paliperidone ER in the fasted state; Treatment B: one 20 mg paroxetine tablet once a day from Day 1 to Day 13 and 1 tablet of 3 mg paliperidone ER on Day 10 in the fasted state. Successive paliperidone ER administrations will be separated by a washout period of at least 14 days and no more than 28 days. Paroxetine is a potent and selective CYP2D6 inhibitor. Inhibitors of CYP2D6 such as paroxetine have been reported to increase the plasma concentrations of antipsychotics such as perphenazine, clozapine, and risperidone. Because paliperidone ER and paroxetine could potentially be used in combination in schizophrenic patients, the potential for a drug-drug interaction between paroxetine and paliperidone ER needs to be explored.The safety and tolerability of the 3 mg tablet of paliperidone ER administered with and without paroxetine to healthy men will be monitored.

Two single oral doses of paliperidone ER 3-mg; 20-mg paroxetine orally once a day for 13 days

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (weight [kg]/height [m2]) of 18 to 30 kg/m2, inclusive
* Extensive metabolizer of CYP2D6. Volunteers whose CYP2D6 genotype is unknown should have been phenotyped before the start of the study using dextromethorphan as a probe (i.e., have a dextromethorphan metabolic ratio <0.02, as determined according to the standard procedures of the study center)
* Have a supine (after 5 minutes rest) blood pressure between 100 and 140 mmHg systolic, inclusive, and 50 and 90 mmHg diastolic, inclusive
* Smokes no more than 10 cigarettes, or 2 cigars, or 2 pipes per day and has been following this pattern for at least 3 months before screening
* Healthy on the basis of a prestudy physical examination, medical history, 12-lead ECG, and the laboratory results of serum chemistry, hematology, and urinalysis performed within 21 days before the first dose. If the results of the serum chemistry, hematology, or urinalysis testing are not within the laboratory's reference ranges, the volunteer can be included only if the investigator judges that the deviations are not clinically significant. For renal function tests, the values must be within the normal laboratory reference ranges

Exclusion Criteria:

* Poor or intermediate metabolizers of CYP2D6, as determined by genotyping or phenotyping using dextromethorphan
* Known drug allergy to risperidone, paliperidone, paroxetine, or any of their excipients
* Known history of drug-induced dystonia
* Recent history of alcohol or substance abuse
* Relevant history or presence of any cardiovascular (including myocardial infarct or cardiac arrhythmia), respiratory, neurologic (including seizures), psychiatric, renal, hepatic, gastrointestinal (including surgeries, severe gastrointestinal narrowing, and malabsorption problems), endocrine, hematologic, or immunologic disease
* History of any cancer, with the exception of basal cell carcinoma
* At screening, has signs of autonomic dysfunction as indicated by a sustained decrease of >20 mmHg in systolic blood pressure or a decrease of >10 mmHg in diastolic blood pressure after standing for at least 2 minutes that is not associated with an increase of >15 beats per minute (bpm) in heart rate
* Bradycardia (heart rate <50 bpm) as determined by screening 12-lead ECG
* A positive test result (or history of) for any of the serology tests (hepatitis B and C, and human immunodeficiency virus) at screening

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2006-03; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the effects of a CYP2D6 inhibitor, paroxetine, on the pharmacokinetics of a single dose of orally administered paliperidone ER

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of the 3 mg tablet of paliperidone ER administered with and without paroxetine to healthy men

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A study of the effects of paroxetine on the pharmacokinetics of paliperidone ER — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=711&filename=CR007561_CSR.pdf